CLINICAL TRIAL: NCT07109011
Title: Feasibility, Acceptability, and Validation of a User-friendly Diet Quality Tool in Adults From Ambulatory Nutrition Clinics: the PLATE Study
Brief Title: Feasibility, Acceptability, and Validation of a User-friendly Diet Quality Tool in Adults From Ambulatory Nutrition Clinics
Acronym: PLATE
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Charlene Compher, Professor, University of Pennsylvania
Other Study IDs: 855371
Record Dates: First submitted 2025-07-25; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Weight Management; Cardiovascular (CV) Risk; Metabolic and Nutritional Disorders
Keywords: diet quality; nutrition counseling; Healthy Eating Index; food photography; validation
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study design for Perceptions and Learning About a Diet Tool (PLATE) was a prospective online dietary intake survey in adults engaged in ambulatory nutrition counseling.

DETAILED DESCRIPTION:
Adults over the age of 18 years who attended a nutrition counseling visit in the health system's outpatient clinics within the past six months and who had agreed to be contacted for potential research participation were eligible. Monthly reports from the electronic health record of patients from nutrition counseling visits were used to identify potential participants. A link to the study consent form and surveys was sent to these patients by email.

ELIGIBILITY:
Inclusion Criteria:

* Adults who attended a nutrition counseling visit at Penn Medicine within past 6 months

Exclusion Criteria:

* No nutrition counseling visit within past 6 months, age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who attended nutrition counseling visit at Penn Medicine within the past 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Acceptability of cellphone photos | 3 days
  survey questions about ease of use of cellphone for photos, comfort sending photos to study team, preference for food photos for diet intake reporting in the future on Likert scale.

SECONDARY OUTCOMES:
Test-retest replicability | 4-10 days
  Diet screening tool, Penn Healthy Diet-Goals (PHD-G), is a 36-item self-report survey of food groups based on Healthy Eating Index and food examples from NHANES. The tool is completed once by the participant independently and then a second time by assistance of study personnel during a phone call4-10 days later.
Validity of Penn Healthy Diet-Goals (PHD-G) survey relative to 3-day food record. | 4-10 days between first food record day and following PHD-G.
  Food groups reported on PHD-G survey will be compared to those reported in the food record.

CONTACTS AND LOCATIONS:
Overall Officials: Charlene W Compher, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD may be shared upon request and approval of the authors.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 7/25/2025-7/24/2026
Access Criteria: Investigators who request permission from the PI for a specific analytical question will be evaluated for potential deidentified data sharing.